CLINICAL TRIAL: NCT03494803
Title: Clinical Trials on Detection of Prostate Cancer With Non-invasive Method Based on DNA Methylation of Circulated Tumor DNA, PBMC and T Cells
Brief Title: Detection of Prostate Cancer With Non-invasive Method Based on DNA Methylation of Circulated Tumor DNA, PBMC
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled, leading to insufficient patient numbers to initiate the clinical trial.
Sponsor: HKGepitherapeutics (Industry)
Collaborators: Kazakh Research Institute of Oncology & Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: HKG-KZ-PRAD-103
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Cancer Metastatic
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control
- Prostate Cancer

SUMMARY:
Prostate cancer is a leading cause of mortality and morbidity.

The purpose of this study is to develop and test non-invasive biomarkers based on methylation changes in PBMC, T-cells and circulated tumor DNA in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: The patient must sign the appropriate approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Pregnant women
* Minors (subjects less than 18 years of age)
* Prisoners
* Patients having other than one cancer
* Subjects unable to consent for themselves
* Symptomatic of acute prostatitis

Ages: 18 Years to 90 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients will be assigned an ID that will be kept confidential according to hospital regulations. IDs will be randomized so that identity will not be revealed except to the approved hospital personnel. Methylation data will be returned to the hospital for follow up of progression of disease and for assessing early prediction of progression of Prostate cancer and will be entered into the data base. Other clinical follow up data will be entered into the electronic data base. All data will be captured in case report form
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
DNA methylation of circulated tumor and PBMC DNA and its Correlation to Development and prediction of prostate cancer | 6 months to 1 year
  We will develop the linear model and a threshold value differentiating breast cancer from control based on the 100 patient training set. The model will be provided to the researchers:
  Methylation score=CG1*b1+CG2*b2+ CG3*b3 + e
  CG1 is the methylation value of the first CG b1 is the regression coefficient for the first CG and e equals the intercept.
  We will develop the regression coefficient and intercept as well as the DNA methylation values for each patient for each CG. We will first compute the polygenic methylation score for each patient. Then based on the computer threshold based on the training cohort will call the samples as prostate cancer or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided